CLINICAL TRIAL: NCT06185270
Title: Effects of Preoperative Frailty Assessed by Short Physical Performance Battery (SPPB) on Short-term Postoperative Recovery Among Gastric Cancer Patients Undergoing Minimally Invasive Distal Gastrectomy
Brief Title: Effects of Preoperative Frailty on Postoperative Recovery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2308-179-1462
Record Dates: First submitted 2023-11-05; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-11

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing minimally invasive distal gastrectomy for early gastric cancer
  Interventions: Diagnostic Test: SPPB

INTERVENTIONS:
Diagnostic Test: SPPB — Short Physical Performance Battery using the automated device (Andantefit)

SUMMARY:
This study aims to evaluate frailty using Short Physical Performance Battery (SPPB) before surgery and find out how frailty affects short-term postoperative recovery after surgery using Quality of Recovery-15 (QOR-15) questionnaire in patients undergoing minimally invasive distal gastrectomy for early gastric cancer.

DETAILED DESCRIPTION:
As the elderly population increases, the evaluation and management of preoperative frailty is becoming important. In patients with frailty, exposure to external stress, such as surgery, can reduce physical function, increase postoperative complication, and raise the risk of death. This study aims to evaluate frailty using an automated device performing SPPB (Andantefit) and find out how frailty affects postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 70 years of age, undergoing minimal invasive (laparoscopic, robot-assisted) distal gastrectomy for early gastric cancer, who can assess short-term postoperative recovery

Exclusion Criteria:

* Patients who have a difficulty in communication
* Patients who have a major medical or mental disease that can affect treatment outcome
* Patients unsuitable for this clinical trail on the opinion of researcher

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over 70 years of age, undergoing minimal invasive (laparoscopic, robot-assisted) distal gastrectomy for early gastric cancer, who can assess short-term postoperative recovery
Sampling Method: Probability Sample
Enrollment: 139 (Estimated)
Dates: Start 2023-12-26 (Estimated); Primary Completion 2024-12-25 (Estimated); Study Completion 2024-12-25 (Estimated)

PRIMARY OUTCOMES:
Poor postoperative outcome (the Korean version of Quality of Recovery-15 [QoR-15K] < 122) | on postoperative day 3
  The minimum and maximum values of QoR-15K are 0 and 150, respectively. Higher scores mean better outcomes.

SECONDARY OUTCOMES:
Poor postoperative outcome (the Korean version of Quality of Recovery-15 [QoR-15K] < 122) | on postoperative day 1
  The minimum and maximum values of QoR-15K are 0 and 150, respectively. Higher scores mean better outcomes.
Poor postoperative outcome (the Korean version of Quality of Recovery-15 [QoR-15K] < 122) | on postoperative day 2
  The minimum and maximum values of QoR-15K are 0 and 150, respectively. Higher scores mean better outcomes.

OTHER OUTCOMES:
Postoperative QoR-15K score | postoperative day 1, 2, 3
  The minimum and maximum values of QoR-15K are 0 and 150, respectively. Higher scores mean better outcomes.
Pain score at rest / during ambulation | postoperative day 1, 2, 3
  Measuring with 11-pointed numeric rating scale (NRS). The minimum and maximum values of NRS are 0 and 11, respectively. Higher score means a more severe pain.
Ambulation distance | postoperative day 1, 2, 3
  Total ambulation distance for a day. Measured by pedometer
First gas out time | up to 1 week after surgery
  Measurement of the time until the first gas out after surgery
Postoperative complication | up to 1 month after surgery
  Based on Clavien-Dindo classification, Grade I-V
Hospital length of stay | at the day of discharge (up to 1 month after admission)
  Measurement of the time until discharge after surgery